CLINICAL TRIAL: NCT06273202
Title: Ultrasound Monitoring of Muscle Thickness in Premature Patients Undergoing Infant Massage: Experience in a Neonatal Intensive Care Unit
Brief Title: Ultrasound Monitoring of Muscle Thickness in Premature Patients
Acronym: NeoMassage
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Policlinico Universitario Agostino Gemelli IRCCS (Other)
Responsible Party: Principal Investigator, Nobile Stefano, Principal investigator, Fondazione Policlinico Universitario Agostino Gemelli IRCCS
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6257
Record Dates: First submitted 2024-02-09; First posted 2024-02-22 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: Prematurity
Keywords: prematurity; Infant Massage; Thigh ultrasound; muscle ultrasound
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Massage (Experimental): Infants will be randomized to receive infant massage or not. Infant massage will be performed three times a day (10 minutes per session) until they reach the 35th week of post-conceptional age (35+6) by the two departmental physical therapists (ADP and ADV).
  Interventions: Other: Infant Massage
- Control group (standard care) (No Intervention): Infants in this group will receive standard care.

INTERVENTIONS:
Other: Infant Massage — Infant massage will be performed three times a day (10 minutes per session) until they reach the 35th week of post-conceptional age (35+6) by the two departmental physical therapists (ADP and ADV).
  Arms: Massage

SUMMARY:
The goal of this interventional study is to investigate through musculoskeletal ultrasonography how the thickness and muscle trophism in infants aged 28 to 35 weeks undergoing infant massage compared with a group of infants with similar characteristics not subjected to treatment.

The main questions it aims to answer are:

* To assess by musculoskeletal ultrasound the impact of infant massage on muscle thickness muscle. Specifically, changes in muscle thickness and trophism of the quadriceps femoris.
* Potential effects on spontaneous motility and stature-ponderal growth of infants. In addition, the discomfort and behavioral status of the infant before and after massage will be investigated infant.

Patients included in the study will be randomized according to a random sequence with a 1:1 ratio into theexperimental group (GS) or the control group (GC). Patients in the GS will perform therapy with infant massage in addition to the usual rehabilitation therapies as specified by the program individual habilitative, to which patients in the control group will be subjected exclusively control.

Infant massage will be performed three times a day (10 minutes per session) until they reach the 35th week of post-conceptional age (35+6) by the two departmental physical therapists (ADP and ADV).

Ultrasound will be performed at the time of randomization (T0) and then 1 time per week until the 35th week by two operators (SN and VA); at the same time, the circumference of the thigh subjected to ultrasound examination. A 12Hz linear ultrasound probe will be used, applied perpendicular to the skin. The infant will be placed supine, with the thigh extended, in a neutral position; excessive compression will be avoided by applying a generous amount of gel. At the midpoint of the thigh, the thickness of the quadriceps muscle will be calculated by measuring the distance between the cortex of the femur and the most superficial muscle fascia. The average of at least 2 measurements will be then calculated. The Heckmatt scale will be used to assess the echogenicity of muscle and bone. In addition, at time T0 and at week 35 the following data will be collected: weeks gestational age, weight at birth and at the end of treatment, rectal temperature, blood gas parameters if present.

ELIGIBILITY:
Inclusion Criteria:

* gestational age between 28and 35 weeks;
* day of life ≥ 7 (to ensure passing the transition phase);
* clinically stable infants, either in spontaneous breathing or ventilatory support invasive or noninvasive, with a good ability to regulate states and good stress management.

Exclusion Criteria:

* Brain pathologies;
* Dysmorphisms;
* Clinically unstable patients requiring treatment with inotropes and/or nitric oxide nitric acid and/or drug therapy for closure of the ductus arteriosus of Botallo.

Ages: 28 Weeks to 35 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Quadriceps femuri thickness | Change of quadriceps femur thickness from baseline at 1, 2,3,4,5 weeks
  Thigh ultrasound will be performed to measure quadriceps femuri thickness
Quadriceps femuri trophism | Change of quadriceps femur tropism from baseline at 1, 2,3,4,5 weeks
  The Heckmatt scale will be used to assess muscle trophism (grades I to IV, where I is normal and IV abnormal)

SECONDARY OUTCOMES:
To valuate the discomfort/behavioral status of the infant. | Change of discomfort ,behavioral status of the infant from baseline at 1, 2,3,4,5 weeks
  Assessment by N-PASS: Neonatal Pain, Agitation and Sedation Scale (0-no pain to 10-pain) Anamnestic collection of information on the child's behavioral status: crying, consolability, adjustment to states, stress response (tidal; tremors; startle); activity level.
To valuate the potential effects on spontaneous motility. | Change of General Movement Optimality Score of the infant from baseline at 1, 2,3,4,5 weeks
  Assessment by Prechtl General Movement Optimality Score, from 5 (worse) to 42 (normal)
To evaluate differences in ponderal growth. | Change of General Movement Optimality Score of the infant from baseline at 1, 2,3,4,5 weeks
  Body weight measurement (grams).

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nobile, MD, PhD, Principal Investigator — Fondazione Policlinico Universitario A. Gemelli, IRCCS
Locations (1):
- Fondazione Policlinico Gemelli IRCCS, Roma, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Bertini G, Elia S, Dani C. Using ultrasound to examine muscle mass in preterm infants at term-equivalent age. Eur J Pediatr. 2021 Feb;180(2):461-468. doi: 10.1007/s00431-020-03846-7. Epub 2020 Oct 20. PMID 33083899
- [Result] Su E, Dalesio N, Pustavoitau A. Point-of-care ultrasound in pediatric anesthesiology and critical care medicine. Can J Anaesth. 2018 Apr;65(4):485-498. doi: 10.1007/s12630-018-1066-6. Epub 2018 Jan 19. PMID 29352416
- [Result] Sitka U. [The startle reaction of the newborn infant]. Zentralbl Gynakol. 1990;112(14):911-9. German. PMID 2264411
- [Result] Neu M, Robinson J. Maternal holding of preterm infants during the early weeks after birth and dyad interaction at six months. J Obstet Gynecol Neonatal Nurs. 2010 Jul-Aug;39(4):401-14. doi: 10.1111/j.1552-6909.2010.01152.x. PMID 20629927
- [Result] Harrison L, Olivet L, Cunningham K, Bodin MB, Hicks C. Effects of gentle human touch on preterm infants: pilot study results. Neonatal Netw. 1996 Mar;15(2):35-42. PMID 8700092
- [Result] Lai MM, D'Acunto G, Guzzetta A, Boyd RN, Rose SE, Fripp J, Finnigan S, Ngenda N, Love P, Whittingham K, Pannek K, Ware RS, Colditz PB. PREMM: preterm early massage by the mother: protocol of a randomised controlled trial of massage therapy in very preterm infants. BMC Pediatr. 2016 Aug 27;16(1):146. doi: 10.1186/s12887-016-0678-7. PMID 27568006
- [Result] Beachy JM. Premature infant massage in the NICU. Neonatal Netw. 2003 May-Jun;22(3):39-45. doi: 10.1891/0730-0832.22.3.39. PMID 12795507
- [Result] Mrljak R, Arnsteg Danielsson A, Hedov G, Garmy P. Effects of Infant Massage: A Systematic Review. Int J Environ Res Public Health. 2022 May 24;19(11):6378. doi: 10.3390/ijerph19116378. PMID 35681968
- [Result] Field T, Diego M, Hernandez-Reif M. Preterm infant massage therapy research: a review. Infant Behav Dev. 2010 Apr;33(2):115-24. doi: 10.1016/j.infbeh.2009.12.004. PMID 20137814
- [Result] Pados BF, McGlothen-Bell K. Benefits of Infant Massage for Infants and Parents in the NICU. Nurs Womens Health. 2019 Jun;23(3):265-271. doi: 10.1016/j.nwh.2019.03.004. Epub 2019 May 3. PMID 31059673
- [Result] Pozzi N, D'Angelo G, Gitto E; Gruppo di Studio Terapia Intensiva della Prima Infanzia della SIN. Why is "early childhood intensive care" an Italian association of neonatology study group? Ital J Pediatr. 2019 Mar 6;45(1):33. doi: 10.1186/s13052-019-0626-x. PMID 30841913
- [Result] van Alfen N, Gijsbertse K, de Korte CL. How useful is muscle ultrasound in the diagnostic workup of neuromuscular diseases? Curr Opin Neurol. 2018 Oct;31(5):568-574. doi: 10.1097/WCO.0000000000000589. PMID 30028736
- [Result] Perri A, Sbordone A, Patti ML, Nobile S, Tirone C, Giordano L, Tana M, D'Andrea V, Priolo F, Serrao F, Riccardi R, Prontera G, Maddaloni C, Lenkowicz J, Boldrini L, Vento G. Early lung ultrasound score to predict noninvasive ventilation needing in neonates from 33 weeks of gestational age: A multicentric study. Pediatr Pulmonol. 2022 Sep;57(9):2227-2236. doi: 10.1002/ppul.26031. Epub 2022 Jun 20. PMID 35670034
- [Result] Dubowitz LM, Dubowitz V, Palmer P, Verghote M. A new approach to the neurological assessment of the preterm and full-term newborn infant. Brain Dev. 1980;2(1):3-14. doi: 10.1016/s0387-7604(80)80003-9. PMID 7416439
- [Result] Einspieler C, Prechtl HF. Prechtl's assessment of general movements: a diagnostic tool for the functional assessment of the young nervous system. Ment Retard Dev Disabil Res Rev. 2005;11(1):61-7. doi: 10.1002/mrdd.20051. PMID 15856440
- [Result] Valla FV, Young DK, Rabilloud M, Periasami U, John M, Baudin F, Vuillerot C, Portefaix A, White D, Ridout JA, Meyer R, Gaillard Le Roux B, Javouhey E, Pathan N. Thigh Ultrasound Monitoring Identifies Decreases in Quadriceps Femoris Thickness as a Frequent Observation in Critically Ill Children. Pediatr Crit Care Med. 2017 Aug;18(8):e339-e347. doi: 10.1097/PCC.0000000000001235. PMID 28650903
- [Result] de Figueiredo RS, Nogueira RJN, Springer AMM, Melro EC, Campos NB, Batalha RE, Brandao MB, de Souza TH. Sarcopenia in critically ill children: A bedside assessment using point-of-care ultrasound and anthropometry. Clin Nutr. 2021 Aug;40(8):4871-4877. doi: 10.1016/j.clnu.2021.07.014. Epub 2021 Jul 21. PMID 34358831
- [Result] Morgan ME, Kukora S, Nemshak M, Shuman CJ. Neonatal Pain, Agitation, and Sedation Scale's use, reliability, and validity: a systematic review. J Perinatol. 2020 Dec;40(12):1753-1763. doi: 10.1038/s41372-020-00840-7. Epub 2020 Oct 2. PMID 33009491
- [Result] Klawitter F, Walter U, Patejdl R, Endler J, Reuter DA, Ehler J. Sonographic Evaluation of Muscle Echogenicity for the Detection of Intensive Care Unit-Acquired Weakness: A Pilot Single-Center Prospective Cohort Study. Diagnostics (Basel). 2022 Jun 2;12(6):1378. doi: 10.3390/diagnostics12061378. PMID 35741188
- [Result] Billingham SA, Whitehead AL, Julious SA. An audit of sample sizes for pilot and feasibility trials being undertaken in the United Kingdom registered in the United Kingdom Clinical Research Network database. BMC Med Res Methodol. 2013 Aug 20;13:104. doi: 10.1186/1471-2288-13-104. PMID 23961782